CLINICAL TRIAL: NCT02065427
Title: Intervention to Improve Social and Family Support for Caregivers of Dependent Patients
Brief Title: Intervention to Improve Social and Family Support for Caregivers of Dependent Patients. (ICIAS)
Acronym: ICIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ICIAS
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Dependency Burden
Keywords: Caregiver; Burden; Social support; Primary health Care; Home Care; Intervention

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social support (Experimental): Social support intervention
  Intervention is performed by the health professionals working at the primary health care team responsible for the patient, and consisits of the following components:
  a) PHCT professionals: standardized training to implement caregivers intervention. b) Caregivers: 1 individualized counselling session, 1 family session, and 4 educational group sessions conducted by participating PHCT professionals; in addition to usual home health care visits, periodic telephone follow-up contact and unlimited telephone support.
  Interventions: Behavioral: Social Support
- Usual home health care (No Intervention): Caregivers and dependent patients: usual home health care, consisting of bimonthly scheduled visits, follow-up as needed, and additional attention upon request

INTERVENTIONS:
Behavioral: Social Support — a) PHCT professionals: standardized training to implement caregivers intervention. b) Caregivers: 1 individualized counselling session, 1 family session, and 4 educational group sessions conducted by participating PHCT professionals; in addition to usual home health care visits, periodic telephone follow-up contact and unlimited telephone support.
  Arms: Social support

SUMMARY:
The purpose of this study is to determine wether a multi-factor intervention involving the primary caregiver of a dependent patient, with the goal of improving his or her social and family support and carried out by the professionals of the patient's regular PHCT, will decrease the burden and increase quality of life for the primary caregiver.

DETAILED DESCRIPTION:
Objective: To assess whether an intervention designed to improve the social support for caregivers effectively decreases caregivers burden and improves their quality of life.

Methodology:

Design: Controlled, multicentre, community intervention trial, with patients and their caregivers randomized to the intervention or control group according to their assigned Primary Health Care Team (PHCT).

Study area: Primary Health Care network (9 PHCTs). Study participants: Primary informal caregivers of patients receiving home health care from participating PHCTs.

Sample: Required sample size is 282 caregivers (141 from PHCTs randomized to the intervention group and 141 from PHCTs randomized to the control group.

Intervention: a) PHCT professionals: standardized training to implement caregivers intervention. b) Caregivers: 1 individualized counselling session, 1 family session, and 4 educational group sessions conducted by participating PHCT professionals; in addition to usual home health care visits, periodic telephone follow-up contact and unlimited telephone support.

Control: Caregivers and dependent patients: usual home health care, consisting of bimonthly scheduled visits, follow-up as needed, and additional attention upon request.

Data Analysis. Dependent variables: Caregiver burden (short-form Zarit test), caregivers social support (Medical Outcomes Study), and caregiver reported quality of life (SF-12) Independent variables: a) Caregiver: sociodemographic data, Goldberg Scale, Apgar family questionnaire, Holmes and Rahe Psychosocial Stress Scale, number of chronic diseases. b) Dependent patient: sociodemographic data, level of dependency (Barthel Index), cognitive impairment (Pfeiffer test)

Discussion:

If the intervention intended to improve social and family support is effective in reducing the burden on primary informal caregivers of dependent patients, this model can be readily applied throughout usual PHCT clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Adults (older than 18 years) identified in the eCAP database as the primary caregiver for a dependent patient, and who act as caregivers without remuneration.

Both the caregivers and the dependent patients have an active clinical record in a participating primary care centre.

-

Exclusion Criteria:

- 1. Caregivers for intermittent periods, independently of the length of care provided.

2. Caregivers who have provided less than one year of ongoing care. 3. Caregivers with any communication problem (psychiatric disorders, etc.) that makes them difficult to interview

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Score in Zarit's short version test for caregiver's burden | 6 months
  Difference in Zarit's score in the primary caregiver for a dependent patient before and after iintervention

SECONDARY OUTCOMES:
Score in caregivers social support (Medical Outcomes Study), (MOS) | 6 months
  Difference in score in MOS Test beefore and after intervention

OTHER OUTCOMES:
Score in caregiver reported quality of life (SF-12) | 6 months
  Diference in score in quality of life ( SF-12 test) before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena I Rosell-Murphy, MD, Study Director — Institut Català de la Salut; Josep Mª Bonet, MD, Principal Investigator — Institut Català de la Salut
Locations (1):
- CAP Rambla, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Rosell-Murphy M, Bonet-Simo JM, Baena E, Prieto G, Bellerino E, Sole F, Rubio M, Krier I, Torres P, Mimoso S; ICIAS research group. Intervention to improve social and family support for caregivers of dependent patients: ICIAS study protocol. BMC Fam Pract. 2014 Mar 25;15:53. doi: 10.1186/1471-2296-15-53. PMID 24666438